CLINICAL TRIAL: NCT01260727
Title: A Phase I Study of the Safety and Immunogenicity of PENNVAX-G DNA (ENV & GAG) Administered by Intramuscular Biojector 2000 or CELLECTRA Intramuscular Electroporation Device Followed by MVA-CMDR (HIV-1 CM235 ENV/CM240 GAG/POL) Boost in Healthy, HIV Uninfected Adults
Brief Title: Evaluating the Safety of and Immune Response to an HIV Vaccine Followed by Booster, Administered by Two Devices, in HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RV 262; 10793 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1 (Experimental): Participants will receive PENNVAX-G vaccine administered by intramuscular injection (IM) via Biojector 2000 needleless device in either deltoid on Days 0 and 28. They will then receive MVA-CMDR administered IM by needle and syringe in either deltoid on Days 84 and 168.
  Interventions: Biological: PENNVAX-G DNA Vaccine; Biological: MVA-CMDR Vaccine
- Group 2 (Experimental): Participants will receive PENNVAX-G vaccine administered via CELLECTRA EP in either deltoid on Days 0 and 28. They will then receive MVA-CMDR administered IM by needle and syringe in either deltoid on Days 84 and 168.
  Interventions: Biological: PENNVAX-G DNA Vaccine; Biological: MVA-CMDR Vaccine
- Group 3: Subgroup 1 (Experimental): Participants will receive PENNVAX-G vaccine administered IM via Biojector 2000 needleless device in either deltoid on Days 0 and 28. They will then receive MVA-CMDR administered IM by needle and syringe in either deltoid on Days 84 and 168.
  Interventions: Biological: PENNVAX-G DNA Vaccine; Biological: MVA-CMDR Vaccine
- Group 3: Subgroup 2 (Placebo Comparator): Participants will receive placebo vaccine for PENNVAX-G administered IM via Biojector 2000 needless device in either deltoid on Days 0 and 28. They will then receive placebo vaccine for MVA-CMDR administered IM by needle and syringe in either deltoid on Days 84 and 168.
  Interventions: Biological: Placebo PENNVAX-G Vaccine; Biological: Placebo MVA-CMDR Vaccine
- Group 4: Subgroup 1 (Experimental): Participants will receive PENNVAX-G vaccine administered IM via CELLECTRA EP in either deltoid on Days 0 and 28. They will then receive MVA-CMDR administered IM by needle and syringe in either deltoid on Days 84 and 168.
  Interventions: Biological: PENNVAX-G DNA Vaccine; Biological: MVA-CMDR Vaccine
- Group 4: Subgroup 2 (Placebo Comparator): Participants will receive placebo vaccine for PENNVAX-G administered IM via CELLECTRA EP in either deltoid on Days 0 and 28. They will then receive placebo vaccine for MVA-CMDR administered IM by needle and syringe in either deltoid on Days 84 and 168.
  Interventions: Biological: Placebo PENNVAX-G Vaccine; Biological: Placebo MVA-CMDR Vaccine

INTERVENTIONS:
Biological: PENNVAX-G DNA Vaccine — PENNVAX-G DNA (HIV-1 env A, C, and D, and consensus gag plasmids) vaccine; 4 mg administered IM as a total volume of 1 mL
  Arms: Group 1; Group 2; Group 3: Subgroup 1; Group 4: Subgroup 1
Biological: MVA-CMDR Vaccine — MVA-CMDR live attenuated modified vaccinia ankara vector (HIV-1 CM235 env/CM240 gag/pol); 1 x 10^8 plaque-forming unit (pfu) administered IM by needle and syringe as a volume of 1 mL in either deltoid
  Arms: Group 1; Group 2; Group 3: Subgroup 1; Group 4: Subgroup 1
Biological: Placebo PENNVAX-G Vaccine — Sodium Chloride Injection USP, 0.9%
  Arms: Group 3: Subgroup 2; Group 4: Subgroup 2
Biological: Placebo MVA-CMDR Vaccine — Sodium Chloride Injection USP, 0.9%
  Arms: Group 3: Subgroup 2; Group 4: Subgroup 2

SUMMARY:
The purpose of this study is to evaluate the safety of and immune response to an HIV vaccine, administered using two different devices, followed by a vaccine boost, in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
Despite advances in treatment, HIV/AIDS rates remain high in low- and middle-income countries in resource-limited areas of the world. Preventive HIV vaccines would be an effective way to decrease the spread of HIV/AIDS. This study will evaluate an experimental HIV preventive vaccine followed by booster: the PENNVAX-G DNA vaccine and the Modified Vaccinia Ankara-Chiang Mai Double Recombinant (MVA-CMDR) booster vaccine. The MVA virus is a mild form of a vaccinia virus that is used in smallpox vaccines and does not cause smallpox infection. It has been safely used in vaccines for many years. Study researchers will examine if the combination of the two vaccines will provide an effective way for the body to build a defense against HIV. The PENNVAX-G vaccine will be administered to participants using one of two devices-the Biojector 2000 needleless device or the CELLECTRA intramuscular (IM) electroporation (EP) device-to evaluate how the immune response to the vaccine changes based on the device that is used. The purpose of this study is to evaluate the safety and immunogenicity of the PENNVAX-G vaccine, administered by either Biojector 2000 injection or CELLECTRA EP, followed by an MVA-CMDR vaccine boost, in healthy, HIV-uninfected adults.

This study will be conducted in two parts. Participants in the first part of the study will attend a baseline study visit, and they will undergo blood and urine collection, a medical history review, physical examination, and HIV testing counseling. All participants will receive the PENNVAX-G vaccine at baseline and Day 28. They will be randomly assigned to receive the vaccine by either the Bioinjector 2000 needleless device or the CELLECTRA IM EP device. On Days 84 and 168, all participants will receive the MVA-CMDR vaccine by IM injection delivered via needle and syringe. Participants will remain in the clinic for 1 hour after each vaccination for observation and vital sign monitoring, and they will record their temperatures and any symptoms in a diary for 7 days after each vaccination. Study staff will contact participants 1 to 2 days after each vaccination for follow-up monitoring. In addition to the vaccination study visits, participants will attend study visits at Weeks 1, 2, 4, 5, 6, 13, 14, 25, 26, 37, 50, and 52 and will repeat the baseline study procedures.

At the conclusion of the first part of the study, participants' study data will be reviewed and the safety of the vaccine regimen will be determined. If the regimen is found to be safe, then the second part of the study will begin. Participants in the second part of the study will be randomly assigned to receive the PENNVAX-G vaccine administered by either the Bioinjector 2000 device or the CELLECTRA EP device at baseline and Day 28, followed by the MVA-CDMR boost at Days 84 and 168, or they will receive placebo PENNVAX-G vaccine administered by either the Bioinjector 2000 device or the CELLECTRA EP device at baseline and Day 28, followed by a placebo MVA-CDMR boost at Days 84 and 168. All study visits and procedures that occurred during the first part of the study will also take place in the second part of the study.

Participants in the second part of the study will have the option of enrolling in a substudy. The purpose of the substudy is to evaluate the antibody response of the reproductive tract mucosa to the PENNVAX-G DNA, MVA-CDMR, and placebo vaccines administered in the main part of study. The substudy will also evaluate the effectiveness of using the Instead Softcup as a collection method to collect vaginal secretions for testing. Mucosal specimens and urine samples will be collected from participants at the screening visit and during the Week 2, 6, 14, 26, and 50 study visits.

ELIGIBILITY:
Inclusion Criteria:

* Low risk of HIV infection (as defined by the Study Risk Assessment Tool captured during the medical history)
* Amenable to HIV risk reduction counseling, committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit, and committed to 18 months of follow-up contact
* Pass the Test of Understanding and demonstrate an understanding of STEP study results (HVTN 502/Merck 023 trial)
* Assessed by the clinic staff as being at low risk of HIV infection on the basis of sexual behaviors within the 12 months prior to enrollment as follows: sexually abstinent, or had two or fewer mutually monogamous relationships with HIV-uninfected partners and who have not used illicit drugs, or had two or fewer partners believed to be HIV uninfected and who did not use illicit drugs and with whom he/she regularly uses condoms for sexual intercourse
* Healthy men and women (determined by medical history, physical examination, and clinical judgment)
* Available and willing to participate for 12 months for study visits and annual follow-up for 18 months after study completion
* Must be willing to have photo or fingerprint taken for identification purposes
* Must be willing to be taken home at enrollment visit and allow home visits, if needed
* Able to read and willing to complete the informed consent process
* Has the following laboratory criteria within 45 days prior to study entry:

  1. Hemoglobin: Women: 11 mg/dL; Men: 12.5 mg/dL
  2. White cell count: 2,500 to 11,000 cells/mm^3
  3. Platelets: 125,000 to 450,000 per mm^3
  4. Urinalysis: protein and blood less than 1+, glucose negative
  5. Normal liver function tests to include alanine aminotransferase (ALT)/aspartate aminotransferase (AST), alkaline phosphatase, gamma-glutamyl transpeptidase (GGT) (less than or equal to 1.25 times the institutional upper limits of normal), creatine phosphokinase (CPK) (less than or equal to 600 IU/L), troponin I (less than 0.4 ng/mL), and creatinine (less than or equal to 1.25 times the institutional upper limits of normal)
  6. Negative for HIV infection (enzyme linked immunosorbent assay [ELISA], Western blot [WB], and HIV polymerase chain reaction [PCR])
* Female participants must have a negative pregnancy test at the screening visit and have a negative pregnancy test immediately prior to each vaccine/placebo vaccination
* Provide verbal assurance that adequate birth control measures have been followed for 45 days prior to the first vaccine/placebo vaccination and will continue to be followed for at least 3 months after the final vaccine/placebo vaccination. More information on this criterion can be found in the protocol.
* Body mass index (BMI) less than 30

Exclusion Criteria:

* Confirmed HIV-1 or HIV-2 infection
* Engaged in excessive daily alcohol use, frequent binge drinking, or illicit drug use within the 12 months prior to study entry
* History of new onset, sexually acquired infection, as determined by local, syndromic diagnostics standards or, as available, serologic and microbiologic diagnosis within the 12 months prior to study entry
* Has a known current high-risk partner or had such a partner within the 12 months prior to study entry
* Hepatitis B, hepatitis C, or syphilis infection; active syphilis documented by exam or serology unless positive serology is because of remote treated infection or positive rapid plasma reagin
* Pregnant, planning on becoming pregnant during the study, or breastfeeding
* Any clinically significant acute or chronic medical condition that, in the opinion of the investigator, would preclude study participation (e.g., history of seizure disorders, bleeding/clotting disorder, autoimmune disease, malignancy, tuberculosis, other systemic infections)
* Major surgery within the 4 weeks prior to study entry
* History of or known active heart disease including:

  1. Previous myocardial infarction (heart attack)
  2. Angina pectoris; congestive heart failure
  3. Valvular heart disease, including mitral valve prolapse
  4. Cardiomyopathy
  5. Myo/pericarditis
  6. Stroke or transient ischemic attack
  7. Chest pain or shortness of breath with activity (such as walking up stairs)
  8. Arrhythmia/episodic palpitations (not excluded: sinus arrhythmia)
  9. Pacemaker
  10. Other heart conditions under the care of a doctor
* People who have the following cardiac risk factors:

  1. Participant report of history of elevated blood cholesterol defined as fasting low-density lipoprotein (LDL) greater than 160 mg/dL
  2. First degree relative (e.g., mother, father, brother, sister) who had coronary artery disease before the age of 50 years
* Electrocardiogram (ECG) with clinically significant findings, or features that would interfere with the assessment of myo/pericarditis. More information on this criterion can be found in the protocol.
* History of diabetes mellitus type 1 or type 2, including cases controlled with diet alone (not excluded: history of isolated gestational diabetes)
* Thyroidectomy or thyroid disease requiring medication during the 12 months prior to study entry
* High blood pressure:

  1. If a person has been diagnosed with high blood pressure during screening or previously, exclude for high blood pressure that is not well controlled. More information on this criterion can be found in the protocol.
  2. If a person has NOT been diagnosed with high blood pressure during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at study entry or diastolic blood pressure greater than or equal to 100 mm Hg at study entry
* Major psychiatric illness and/or substance abuse problems during the 12 months before study entry that, in the opinion of the investigator, would preclude study participation
* Receipt of live attenuated vaccine within 30 days or inactivated/killed vaccine within 2 weeks of DNA vaccination
* Use of experimental therapeutic agents within 30 days of study entry
* Current or planned participation in another clinical study during the study period
* Receipt of blood products or immunoglobulin in the 3 months before study entry
* History of anaphylaxis or other serious adverse reactions to vaccines or egg products or amide type anesthetics (e.g., bupivacaine, novocaine, lidocaine, mepivacaine, neomycin, streptomycin)
* History of chronic urticaria (recurrent hives)
* Chronic or recurrent use of medications that modify host immune response (e.g., cancer chemotherapeutic agents, parenteral corticosteroids [topical not an exclusion])
* Recipient of an HIV vaccine candidate at any time and receipt of other experimental vaccine(s) within the 5 years before study entry. More information on this criterion can be found in the protocol.
* A study site employee
* Military personnel (will be excluded from participation in this study at all sites due to the potential for a false-positive HIV test result on mandatory HIV testing, which could have adverse affects on deployment status)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2010-02; Primary Completion 2013-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Severe local toxicity at injection site | Measured after each vaccination
Severe systemic symptoms judged to be probably or definitely related to the vaccine | Measured after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: MAJ Julie Ake, MD, Study Chair — U.S. Military HIV Research Program (MHRP)/Walter Reed Army Institute of Research (WRAIR)
Locations (4):
- Rockville Vaccine Assessment Clinic (RVAC), Rockville, Maryland, United States
- Kenya Med. Research Inst./Walter Reed Project, Clinical Research Centre, Off Hospital Road. Kericho, Kericho, Kenya
- National Institute for Medical Research (NIMR) - Mbeya Medical Research Center (MMRC) CRS, Mbeya, Tanzania
- Makerere University Walter Reed Project (MUWRP), Kampala, Uganda

REFERENCES:
- [Background] Cristillo AD, Weiss D, Hudacik L, Restrepo S, Galmin L, Suschak J, Draghia-Akli R, Markham P, Pal R. Persistent antibody and T cell responses induced by HIV-1 DNA vaccine delivered by electroporation. Biochem Biophys Res Commun. 2008 Feb 1;366(1):29-35. doi: 10.1016/j.bbrc.2007.11.052. Epub 2007 Nov 26. PMID 18036339
- [Background] Loutfy MR, Harris M, Raboud JM, Antoniou T, Kovacs C, Shen S, Dufresne S, Smaill F, Rouleau D, Rachlis A, Gough K, Lalonde R, Tsoukas C, Trottier B, Walmsley SL, Montaner JS. A large prospective study assessing injection site reactions, quality of life and preference in patients using the Biojector vs standard needles for enfuvirtide administration. HIV Med. 2007 Oct;8(7):427-32. doi: 10.1111/j.1468-1293.2007.00489.x. PMID 17760734
- [Derived] Ake JA, Schuetz A, Pegu P, Wieczorek L, Eller MA, Kibuuka H, Sawe F, Maboko L, Polonis V, Karasavva N, Weiner D, Sekiziyivu A, Kosgei J, Missanga M, Kroidl A, Mann P, Ratto-Kim S, Anne Eller L, Earl P, Moss B, Dorsey-Spitz J, Milazzo M, Laissa Ouedraogo G, Rizvi F, Yan J, Khan AS, Peel S, Sardesai NY, Michael NL, Ngauy V, Marovich M, Robb ML. Safety and Immunogenicity of PENNVAX-G DNA Prime Administered by Biojector 2000 or CELLECTRA Electroporation Device With Modified Vaccinia Ankara-CMDR Boost. J Infect Dis. 2017 Nov 27;216(9):1080-1090. doi: 10.1093/infdis/jix456. PMID 28968759